CLINICAL TRIAL: NCT05549011
Title: Comparison of the Effect of Pericapsular Nerve Group Block and Suprainguinal Fascia Iliaca Compartment Block for Preventing Positioning Pain During Spinal Anesthesia in Orthopedic Hip Surgery Patients: A Prospective Observational Study
Brief Title: PENG vs SIFI Block for Positioning Pain During Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Onur Okur, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 326
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Hip Fractures; Acute Post Operative Pain; Nerve Block; Spinal Anesthesia
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PENG block: This cohort will include participants to whom a PENG block is performed before positioning for spinal anesthesia
  Interventions: Other: PENG Block; Diagnostic Test: Numeric Rating Scale; Diagnostic Test: Angle of sitting
- SIFI block: This cohort will include participants to whom a SIFI compartment block is performed before positioning for spinal anesthesia
  Interventions: Other: SIFI compartment block; Diagnostic Test: Numeric Rating Scale; Diagnostic Test: Angle of sitting

INTERVENTIONS:
Other: PENG Block — PENG block for analgesic purposes performed before hip surgery
  Groups: PENG block
Other: SIFI compartment block — SIFI compartment block for analgesic purposes performed before hip surgery
  Groups: SIFI block
Diagnostic Test: Numeric Rating Scale — Self-reported pain intensity score between 0-10
Diagnostic Test: Angle of sitting — Measurement of sitting angle in degrees with a protractor

SUMMARY:
This study aims to compare the effectiveness of preoperative ultrasound-guided suprainguinal fascia iliaca compartment block (SFICB) and pericapsular nerve group block (PENG) in preventing positioning pain during spinal anesthesia in patients who are scheduled for surgery due to hip fracture.

DETAILED DESCRIPTION:
Patients to whom an analgesic block was placed (either PENG or SIFI compartment analgesic block) to ameliorate positioning pain during spinal anesthesia for hip fracture surgery will be enrolled after written consent is obtained. Patients will be asked to report their pain intensity while sitting and their sitting angle will be measured. Patients will be observed for any possible complications( LAST, allergic reactions, hypotension, bradycardia). Pain intensity will then again be questioned postoperatively along with analgesic consumption at the 24th hour. Patients will be arranged into two cohorts according to the block (PENG vs SIFI) and the data obtained will be compared between two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a hip fracture
* who were scheduled to undergo surgery with spinal anesthetics
* has no neurologic disorders that impair cooperation (e.g dementia)
* has no true allergies to local anesthetics
* has no contraindications for regional or neuraxial anesthesia (e.g bleeding diathesis, severe aortic stenosis)

Exclusion Criteria:

* Childer under the age of 18
* patients scheduled to undergo surgery with general anesthetics
* refusing to participate
* allergies to local anesthetics
* any neurologic disorder that impairs patient cooperation
* any contraindication to regional or neuraxial anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a population of patients in a tertiary medical care center who are scheduled to undergo hip fracture surgery with spinal anesthetics and to whom either of the analgesic blocks PENG or SIFI compartment block is placed.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Positioning pain during spinal anesthesia with 10-point numeric rating scale (NRS) | 30 minutes after the block is placed
  NRS is a self-reported pain scale where patient defines intensity of their pain on a scale of 0 to 10. Zero means the patient has no pain while ten means the patient is experiencing the worst pain possible

SECONDARY OUTCOMES:
Sitting angle during positioning | 30 minutes after the block is placed
  Angle of sitting in degrees measured with a protractor during sitting for spinal anesthesia
Postoperative pain with 10-point numeric rating scale (NRS) | Postoperative day 1
  NRS is a self-reported pain scale where patient defines intensity of their pain on a scale of 0 to 10. Zero means the patient has no pain while ten means the patient is experiencing the worst pain possible

CONTACTS AND LOCATIONS:
Overall Officials: Onur OKUR, Principal Investigator — Prof. Dr. Cemil Taşcıoğlu City Hospital; Müslüm AKKILIC, Study Director — Prof. Dr. Cemil Taşcıoğlu City Hospital
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)